CLINICAL TRIAL: NCT02314091
Title: Long Term Results of Randomized Prospective Comparison of Onlay and Sublay Mesh Repair Techniques for Incisional Hernia
Acronym: IH01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, barış sevinç, M.D., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KonyaTRH
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Onlay (Experimental): Onlay mesh repair group
  Interventions: Procedure: onlay mesh hernioplasty
- sublay (Experimental): Sublay mesh repair group
  Interventions: Procedure: onlay mesh hernioplasty

INTERVENTIONS:
Procedure: onlay mesh hernioplasty

SUMMARY:
Randomised prospective comparison of onlay and sublay mesh repair techniques in incisional hernia

ELIGIBILITY:
Inclusion Criteria:

* Incisional hernia
* Acceptance of the trial

Exclusion Criteria:

* BMI>40
* ASA score of 4
* Severe pulmonary or cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
recurrence | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)